CLINICAL TRIAL: NCT05889585
Title: Morbidity, Long-term Side Effects and Quality of Life in Germ-cell Tumor Long Survivors Treated with High-dose Chemotherapy and Autologous Stem Cell Transplant
Acronym: HGT-QoL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-A00855-36; 2020/3139 (Other: CSET Number)
Record Dates: First submitted 2022-09-30; First posted 2023-06-05 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Germ Cell Tumor
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- high-dose of chemotherapy with autologous transplant and relapse-free after a minimum of 3 years. (Other): Men with a histologically-confirmed (or high level serum tumor marker-based) diagnosis of germ-cell tumor, treated for relapse with high-dose of chemotherapy (HDCT) with autologous transplant at Gustave Roussy and relapse-free after a minimum of 3 years.
  Interventions: Other: quality of life questionnaire
- Treated by orchidectomy only and no evidence of relapse after a minimum of 3 years (Other): Men with a histologically confirmed (or high level serum tumor marker-based) stage I germ cell tumor, treated by orchidectomy only and no evidence of relapse after a minimum of 3 years.
  Interventions: Other: quality of life questionnaire
- Treated by first line cisplatin-based chemotherapy and relapse-free after a minimum of 3 years. (Other): Men with a histologically confirmed (or high level serum tumor marker-based) germ cell tumor and good or intermediate prognosis metastatic disease according to the International Germ-Cell Cancer Collaborative Group (IGCCCG), treated by first line cisplatin-based chemotherapy (and surgery of residual masses if needed), with no evidence of relapse after a minimum of 3 years.
  Interventions: Other: quality of life questionnaire

INTERVENTIONS:
Other: quality of life questionnaire — EORTC-QLQ C-30 questionnaire The Impact of Events Scale (IES-R) Multi-Dimensional Fatigue Inventory The EORTC-QLQ C-30 Vers. 3

SUMMARY:
Intensified chemotherapy is an effective treatment in 30-70% of patients with refractory germ cell tumor. Since most cases are diagnosed before the age of 40, survivors can expect to live another 30 to 50 years after being successfully treated. Long-term side effects and physical and emotional consequences can therefore have a significant impact on daily life. To date, no data of this type is available in France. This study will help clinicians better understand the long-term consequences for relapsed patients receiving high-dose chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at diagnosis
* Treated between 1990 and 2015
* Histologically confirmed diagnosis of germ cell tumor (or high level serum tumor marker-based) and:

Treated for relapse with high-dose of chemotherapy (HDCT) with autologous transplant at Gustave Roussy and relapse-free.

Or Treated by orchiectomy only and no evidence of relapse after a minimum of 3 years.

Or Good or intermediate prognosis metastatic disease according to the IGCCCG, treated by first line cisplatin-based chemotherapy at Gustave Roussy (and surgery of residual masses if needed), with no evidence of relapse.

* Ability to comply with the protocol procedures
* Patient affiliated to a social security system or beneficiary of the same. 6-Who have signed a written informed consent form prior to any study specific procedure.

Exclusion Criteria:

* Diagnosis of second malignancy
* Any other serious or unstable illness, or medical, social, or psychological condition, that could jeopardize the safety of the subject and/or his compliance with study procedures, or may interfere with the subject's participation in the study or evaluation of the study results.
* Patient under guardianship or deprived of his/her liberty by a judicial or administrative decision, or incapable of giving his/her consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Compare the quality of life between the three groups measured with the EORTC-QLQ C-30 questionnaire. | Day 1
  To compare the quality of life in long-term survivors of germ cell cancers after high-dose chemotherapy and autologous stem cell transplant with a group of coetaneous patients treated by orchidectomy only for localized testicular tumor and a group of patients of the same age treated with first line cisplatin-based chemotherapy for good or intermediate prognosis advanced germ cell tumor.

SECONDARY OUTCOMES:
Compare late side effects between the three groups. | Day 1
Compare correlated morbidities between the three groups. | Day 1
Compare fatigue measured by the MFI-20 scale between the three groups. | Day 1
Compare symptoms of post-traumatic stress measured by the IES scale between the three groups. | Day 1
Compare current social and professional situation between the three groups. | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, France